CLINICAL TRIAL: NCT00066729
Title: A Phase I Study Of NY-ESO-1b Peptide Plus Montanide ® ISA-51 In Patients With Ovarian, Primary Peritoneal, Or Fallopian Tube Cancer
Brief Title: Vaccine Therapy in Treating Patients With Ovarian Epithelial, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000318803; MSKCC-03034 (Other: Memorial Sloan-Kettering Cancer Center); LUD2002-014 (Other: Ludwig Institute for Cancer Research)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; primary peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NY-ESO-1b peptide with Montanide® ISA-51 (Experimental): Patients received NY-ESO-1b peptide mixed with Montanide® ISA-51 by subcutaneous injections, once every 3 weeks (weeks 1, 4, 7, 10, and 13) for a total of 13 weeks.
  Interventions: Biological: NY-ESO-1 peptide vaccine

INTERVENTIONS:
Biological: NY-ESO-1 peptide vaccine — NY-ESO-1b peptide 100 μg mixed with 0.5 mL of Montanide® ISA-51

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: A phase I trial to study the side effects of vaccine therapy in patients with ovarian epithelial, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of NY-ESO-1b peptide vaccine and Montanide® ISA-51 in patients with ovarian epithelial, primary peritoneal, or fallopian tube cancer.
* Determine the immunologic profile (NY-ESO-1 antibody, CD8+ cells, and delayed-type hypersensitivity) induced by this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive NY-ESO-1b peptide vaccine emulsified with Montanide® ISA-51 subcutaneously once every 3 weeks on weeks 1, 4, 7, 10, and 13 in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 weeks (week 16) and then every 6-12 weeks for 2 years or until disease progression.

ELIGIBILITY:
Inclusion Criteria

1. Histologically documented epithelial carcinoma arising in the ovary, fallopian tube, or peritoneum, from Stage II-IV at diagnosis, receiving initial cytoreductive surgery and chemotherapy with at least one platinum-based chemotherapy regimen.
2. High risk feature defined as suboptimal primary debulking (remaining tumor masses with diameter ≥ 1.0 cm) or failure to normalize CA125 during primary therapy by the end of the third cycle or positive second-look surgery.
3. Patients must be in complete clinical remission defined as CA125 < 35 units, negative physical examination and no definite evidence of disease by computed tomography (CT) of the abdomen and pelvis. Lymph nodes and/or soft tissue abnormalities ≤ 1.0 cm that are often present in the pelvis may not be considered definite evidence of disease.
4. Expected survival of at least 6 months.
5. Karnofsky performance scale ≥60%.
6. Within the last 2 weeks prior to study day 1, vital laboratory parameters should be within normal range, except for the following laboratory parameters, which should be within the ranges specified:

   * Absolute neutrophil count (ANC) ≥1000/mm^3
   * Platelets ≥ 80,000/mm^3
   * Creatinine ≤ 1.5mg/dL
   * Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), and total bilirubin all < 2.5 x upper limit of normal (ULN) 7 Age ≥ 18 years.

8. Able and willing to give valid written informed consent. 9. HLA A02 positive. Exclusion Criteria

Patients were excluded from the study for any of the following reasons:

1. Clinically significant heart disease (NYHA Class III or IV).
2. Other serious illnesses, e.g., serious infections requiring antibiotics or bleeding disorders.
3. Patients with serious intercurrent illness, requiring hospitalization.
4. Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available.
5. Patients taking immunosuppressive drugs such as systemic corticosteroids or non-steroidal anti-inflammatory drugs.
6. Known HIV positivity.
7. Other malignancy within 3 years prior to entry into the study, except for treated nonmelanoma skin cancer and cervical carcinoma in situ.
8. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
9. Lack of availability for immunological and clinical follow-up assessments.
10. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
11. Pregnancy or breastfeeding.
12. Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2003-06-23 (Actual); Primary Completion 2006-05-09 (Actual); Study Completion 2013-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Dupont, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diefenbach CS, Gnjatic S, Sabbatini P, Aghajanian C, Hensley ML, Spriggs DR, Iasonos A, Lee H, Dupont B, Pezzulli S, Jungbluth AA, Old LJ, Dupont J. Safety and immunogenicity study of NY-ESO-1b peptide and montanide ISA-51 vaccination of patients with epithelial ovarian cancer in high-risk first remission. Clin Cancer Res. 2008 May 1;14(9):2740-8. doi: 10.1158/1078-0432.CCR-07-4619. PMID 18451240

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NY-ESO-1b Peptide With Montanide® ISA-51
Started | 9
Completed | 7
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Population: All patients entered into the study.
Arm/Group | NY-ESO-1b Peptide With Montanide® ISA-51
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
NY-ESO-1 Tumor Expression [Count of Participants; unit: Participants]
  Positive | 4
  Negative | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLTs)
Description: Toxicities and adverse events defined by National Cancer Institute Common Toxicity Criteria (CTC) Scale (Version 2.0, published April 30, 1999). DLT defined as:
  ≥ Grade 2 autoimmune phenomena, asymptomatic bronchospasm or generalized urticaria, or ≥ Grade 3 hematological and non hematological toxicities. To be dose-limiting, an adverse event must be definitely, probably, or possibly related to the administration of the investigational agent.
Time Frame: up to 16 weeks
Population: All patients who entered the study and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1b Peptide With Montanide® ISA-51
Number analyzed (Participants) | 9
Participants | 0

2. Secondary Outcome: Number of Patients Developing NY-ESO-1 Antibodies After Treatment
Description: Blood samples were obtained at baseline and in weeks 4, 7, 10, 13 and 16 for the assessment of NY-ESO-1 specific antibodies by enzyme-linked immunosorbent assay (ELISA).
Time Frame: up to 16 weeks
Population: All patients who entered the study and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1b Peptide With Montanide® ISA-51
Number analyzed (Participants) | 9
Participants
  Number of Patients with NY-ESO-1 Antibodies Before and After Treatment | 2
  Number of Patients with No NY-ESO-1 Antibodies Before and After Treatment | 7

3. Secondary Outcome: Number of Patients With NY-ESO-1b-Specific CD8+ T Cells Measured by Tetramer Analysis
Description: Blood samples were obtained at baseline and at 4, 7, 10. 13 and 16 weeks. Tetramer assays were conducted after presensitization of CD8+ T cells with NY-ESO-1b. Results are presented separately for patients with NY-ESO-1 positive and negative tumors.
Time Frame: up to 16 weeks.
Population: All patients who entered the study and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1b Peptide With Montanide® ISA-51
Number analyzed (Participants) | 9
Participants
  Patients with NY ESO-1 Positive Tumors: number analyzed (Participants) | 4
  Patients with NY ESO-1 Positive Tumors: CD8+ T cell immunity by positive tetramer | 3
  Patients with NY ESO-1 Positive Tumors: No CD8+ T cell immunity by tetramer analysis | 1
  Patients with NY-ESO-1 Negative Tumors: number analyzed (Participants) | 5
  Patients with NY-ESO-1 Negative Tumors: CD8+ T cell immunity by positive tetramer | 3
  Patients with NY-ESO-1 Negative Tumors: No CD8+ T cell immunity by tetramer analysis | 2

4. Secondary Outcome: Number of Patients With NY-ESO-1b-Specific Activated CD8+ T Cells Measured by ELISPOT
Description: Blood samples were obtained at baseline and at 4, 7, 10, 13 and 16 weeks. T cell responses were monitored after the in vitro sensitization with NY-ESO-1b (157-165), modified NY-ESO-1b-A (157-165A), or control peptide influenza matrix 58 to 66. Results are presented separately for patients with NY-ESO-1 positive and negative tumors.
Time Frame: up to 16 weeks
Population: All patients who entered the study and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1b Peptide With Montanide® ISA-51
Number analyzed (Participants) | 9
Participants
  Patients with NY-ESO-1 Positive Tumors: number analyzed (Participants) | 4
  Patients with NY-ESO-1 Positive Tumors: Number of patients with CD8+ T cell immunity | 3
  Patients with NY-ESO-1 Positive Tumors: Number of patients without CD8+ T cell immunity | 1
  Patients with NY-ESO-1 Negative Tumors: number analyzed (Participants) | 5
  Patients with NY-ESO-1 Negative Tumors: Number of patients with CD8+ T cell immunity | 3
  Patients with NY-ESO-1 Negative Tumors: Number of patients without CD8+ T cell immunity | 2

5. Secondary Outcome: Number of Patients With NY-ESO-1b-specific Delayed-type Hypersensitivity (DTH)
Description: NY-ESO-1b-specific delayed-type hypersensitivity (DTH) was measured by number of patients with induration and/or redness at each timepoint.
  NY-ESO-1b-specific DTH skin reaction was measured at baseline and weeks 7 and 16. The NY-ESO-1b peptide solution (0.1 mg/mL in 8% DMSO) was injected intradermally at a separate site from the vaccination to give a visable and palpable skin depot. The extent and intensity of DTH reactions were documented by measuring visible redness, palpable induration and other signs of local skin irritation or necrosis. Assessment of DTH reaction was performed 48 hours after injection, and the diameter of the reaction was documented.
Time Frame: up to 16 weeks
Population: All patients who entered the study, received treatment and had at least 1 post-baseline DTH test.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1b Peptide With Montanide® ISA-51
Number analyzed (Participants) | 9
Participants
  DTH Reaction | 0
  No DTH Reaction | 9

6. Post Hoc Outcome: Clinical Outcome as Measured by Number of Patients With No Evidence of Disease and Number of Participants Who Progressed
Description: Although clinical outcome was not an endpoint of this study, patients were evaluated for disease progression throughout the study by cancer antigen 125 (CA-125) levels, physical examination and at the time of study completion with CT scan. All patients enrolled in the study were confirmed to be in Complete Response (cCR) at the initiation of therapy, as documented by CA-125 at <35 units/mL, physical examination, and CT scan without evidence of disease. Patients were assessed for disease progression by CA-125 during the study at weeks 7 and 16. CT scan was done after completion of the study (week 16). After completion of the study, patients returned to the care of their primary treating oncologist, and monitoring was at the discretion of the treating physician.
  No evidence of disease (NED) was defined as no consistent increase in CA-125 or evidence of new lesions on CT scans. Progression was defined as the appearance of new lesions on CT scan.
Time Frame: up to 52 months
Population: All patients who entered the study and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NY-ESO-1b Peptide With Montanide® ISA-51
Number analyzed (Participants) | 9
Participants
  Week 16 (End of Study): NED | 7
  Week 16 (End of Study): Progression | 2
  Month 52 (last follow-up): NED | 3
  Month 52 (last follow-up): Progression | 6

ADVERSE EVENTS:
Time Frame: up to 16 weeks
Description: All Adverse Events (AEs) occurring during the study were to be documented in the source records and on the respective AE Case Report Form (CRF), regardless of the assumption of a causal relationship. All events, which occurred after signed informed consent, were to be documented. All adverse events were graded according to the National Cancer Institute Common Toxicity Criteria (CTC) Scale (Version 2.0, published April 30, 1999).
Arm/Group | NY-ESO-1b Peptide With Montanide® ISA-51
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NY-ESO-1b Peptide With Montanide® ISA-51 (N=9)
Alkaline phosphatase (Investigations) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Abdominal hernia (Gastrointestinal disorders) | 1
Alanine aminotransferase (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin (Investigations) | 3
Blood magnesium decreased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Breath odor (Gastrointestinal disorders) | 1
Catheter site erythema (General disorders) | 1
Confusional state (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Coordination abnormal (Nervous system disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Dyspnea (Cardiac disorders) | 1
Fatigue (General disorders) | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Hemoglobin (Investigations) | 4
Hot flush (Reproductive system and breast disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypothyroidism (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neuropathy (Nervous system disorders) | 4
Neutrophil count (Investigations) | 5
Phootpsia (Eye disorders) | 1
Platelet count (Investigations) | 2
Prothrombin time (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin exfloliation (Skin and subcutaneous tissue disorders) | 1
Syncope (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight increased (Investigations) | 1
White blood cell count (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No